CLINICAL TRIAL: NCT06207851
Title: A Single-arm, Single-center, Open-label, Pilot Clinical Study to Evaluate the Efficacy and Safety of Transcatheter Arterial Micro-Embolization (TAME) Using Nexsphere-F in Patients With Chronic Pain in Elbow or Wrist
Brief Title: Transcatheter Arterial Micro-Embolization (TAME) Using Nexsphere-F in Patients With Chronic Pain in Elbow or Wrist
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS-F TAME002
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): If abnormal blood vessels related to pain are identified by angiography, selective embolization is performed using Nexsphere-F.
  Interventions: Device: Transcatheter Arterial Micro-Embolization

INTERVENTIONS:
Device: Transcatheter Arterial Micro-Embolization — Participants will undergo TAME with Nexsphere-F.

SUMMARY:
In patients with chronic elbow or wrist pain, the pain is controlled by conventional conservative therapy The pain reduction effect of Nexsphere-F embolization in patients who need additional treatment It is intended to demonstrate safety.

DETAILED DESCRIPTION:
This clinical trial is a single cancer, single center, open label, and pilot clinical trial that demonstrates the performance and safety of Nexsphere-F for patients aged 19 to 80 who need additional treatment because their pain is not controlled even after taking existing treatments.

In addition, through this clinical trial, complications of embolization and Nexsphere-F and It checks the safety of side effects. Therefore, in this study, TAME treatment for patients with chronic elbow pain 2 to 7 months, 1 month later, 3 months, 6 wah VAS score reductions and QuickDASH scores, PRTEE score primary 6 Evaluate the reduction rate of medication, discontinuation rate of combination therapy, and occurrence of abnormal cases during the follow-up period. For patients with chronic wrist pain, VAS score after 2 to 7 days, 1 month, 3 months, and 6 months of TAME treatment QuickDASH score reduction rate, drug reduction rate after 6 months, discontinuation rate of combination therapy, and follow-up period the investigators will evaluate the effectiveness and safety of Nexsphere-F by evaluating whether abnormal cases occur during the period.

ELIGIBILITY:
Inclusion Criteria:

1. Those aged 19 to 80
2. Anyone who can provide a consent form
3. A person with a life expectancy of at least 12 months
4. Those who have not responded or failed in preservation treatment for at least three months(e.g. NSAIDS/physical therapy/steroidal joint injections, etc.)
5. VAS score of 4 or higher and moderate-severe elbow or wrist pain

Exclusion Criteria:

1. Those with a VAS Score of less than 4 and Mild Elbow or Wrist Pain
2. Chronic Renal Insufficiency(Serum creatinine > 2mg/dL)
3. allergy to iodide contrast agents that do not respond to steroids
4. Those with acute infection or malignancy
5. Those who have previously had elbow or wrist surgery
6. Those with Bleeding Diabetes that cannot be calibrated

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-07-13 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects with a 50% or more reduction in QuickDASH Score Change | 2~7days,1 month, 3 months, 6 months
  Descriptive statistics (mean, standard deviation, median, minimum and maximum) are presented for each visit compared to the average change rate baseline of the QuickDASH score before and after clinical trial medical device application.

SECONDARY OUTCOMES:
Rate of VAS Score (patient pain intensity) Change | 2~7days,1 month, 3 months, 6 months
  The rate of change of VAS Score (patient pain intensity)Score before and after application of medical devices for clinical trials.(The visual analog scale(VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain." (10). The ends are defined as the extreme limits of the parameter to be measured(symptom,pain,health) orientated from the left(0, worst) to the right(10, best).)
Rate of Changes in symptoms according to in QuickDASH Score | 2~7days,1 month, 3 months, 6 months
  The rate of change of QuickDASH Score before and after application of medical devices for clinical trials.(Change in Patient-Reported Function as measured by the short form Disabilities of the Arm, Shoulder, and Hand (QuickDASH) questionnaires. QuickDASH scores range from 0 (no disability) to 100 (most severe disability.))
Rate of Changes in symptoms according to the Patient-Rated Tennis Elbow Evaluation (PRTEE) Score | 2~7days,1 month, 3 months, 6 months
  The rate of change of Patient-Rated Tennis Elbow Evaluation (PRTEE) Score before and after application of medical devices for clinical trials.((Measurements the patient functional status its 15 questionnaires In PRTEE First subscale is The Pain Subscale detail is 5 items Maximum or best score is 0 and worst score is 50 The Second Subscale or PRTEE is The Specific Activities detail is 6 items with finest score is 0 and least score is 60 The third one subscale of PRTEE the Usual Activities sub part 4 items with superior score is 0 and least score is 40. Third Fourth Part of PRTEE is The Function Subscale detail is performance bases specific activities and usual or regular activities Add up to specific or regular activities divided by 2 Maximum best score or prime score is 0 and least score is 50 Total detail Score of PRTEE is = Pain Subscale + Function Subscale Best Score= 0 Worst Score = 100 (pain and disability contribute equally to score).)
The rate of reduction of medication | 6 months
  The rate of change of medication before and after application of medical devices for clinical trials.

OTHER OUTCOMES:
Number of participants with abnormal cases during follow-up | 1day ,2~7days,1 month, 3 months, 6 months
  Abnormal cases that occurred after the application of medical devices for clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: Sang Woo Park, Principal Investigator — Konkuk Hospital
Locations (1):
- Konkuk Hospital, Seoul, Kwang Jin Gu, South Korea